CLINICAL TRIAL: NCT04559113
Title: Perks of Methylprednisolone for Hospitalized COVID-19 Patients: A Clinical Trial
Brief Title: Methylprednisolone in COVID-19 Patients (Methyl19LGH)
Acronym: Methyl19LGH
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Lahore General Hospital (Other Government)
Responsible Party: Principal Investigator, Dr. M.Irfan Malik, Associate Professor of Pulmonology / Focal Person COVID-19, Lahore General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LGH005
Record Dates: First submitted 2020-09-15; First posted 2020-09-22 (Actual); Last update posted 2020-12-08 (Actual); Status verified 2020-12

CONDITIONS: SARS-CoV Infection; SARS (Severe Acute Respiratory Syndrome)
Keywords: COVID-19; Methylprednisolone; Clinical outcome
MeSH Terms: conditions — Severe Acute Respiratory Syndrome; COVID-19

STUDY DESIGN:
Intervention Model Description: quasi-experimental
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Group intervene with Methylprednisolone (Experimental): Review effect of Methylprednisolone as clinical trial among hospitalized patients with COVID-19 infection.
  Anyone of the following Corticosteroids dose will be given to moderate disease patients of COVID-19
  1. 0.5mg to 1mg/Kg methylprednisolone or equivalent dexamethasone dose (to a maximum of 20mg) given daily x 5 to 7-days or
  2. Methylprednisolone 1 mg/kg daily IV for 5 days followed by 40 mg daily x 3 days, followed by 10 mg daily x 2 day. *Note: in Diabetic patients' dose of methyl prednisolone should be divided in doses preferably 40mg BD.
  Interventions: Drug: Methylprednisolone Injectable Product

INTERVENTIONS:
Drug: Methylprednisolone Injectable Product — 1. 0.5mg to 1mg/Kg methylprednisolone or equivalent dexamethasone dose (to a maximum of 20mg) given daily x 5 to 7-days or
  2. Methylprednisolone 1 mg/kg daily IV for 5 days followed by 40 mg daily x 3 days, followed by 10 mg daily x 2 day.
  Other Names: solu madrol

SUMMARY:
In COVID-19 deep airway and alveolar destruction occurred due to inflammatory reaction resulting into severe pneumonia. In COVID-19, lung injury is not only due to viral damage to tissue, but it is also due to immune response that leads to activation of inflammatory cells and release of cytokines. In COVID-19 acute respiratory distress syndrome ARDS is produced due to mucinous or cellular fibromyxoid exudates, desquamation of pneumocytes and alveolar damage and hyaline membrane development and within 5-7 days disease become more aggressive due to pneumonia and respiratory failure. It is important to start the prompt and strengthen treatment for suppression of inflammatory response and cytokine storm. Methylprednisolone are the traditional immunosuppressive drugs. They are important and effective to delay the pneumonia progression and treating the ARDS.

Corticosteroids are broadly used as treatment for ARDS and there was an evidence for its efficacy for treating SARS and decreasing mortality of SARS in the past. However for COVID-19 corticosteroids efficacy and safety usage is still under clinical trials

DETAILED DESCRIPTION:
All new decision and new interventions that are made for decreasing dependency of ventilator in patients and decreasing patients mortality would have played a great role on global public health. The aim of the study is to address the efficacy of methlyprednisolone for the treatment of COVID-19 patients and its clinical outcome at a tertriary care hospital.

ELIGIBILITY:
Inclusion Criteria:

* All patients of all ages, males, and females who will be diagnosed COVID-19 positive by RT-PCR with moderate illness.
* Patients having classical radiological lesions of COVID-19 on X-ray chest or HRCT chest.
* Respiratory rate > 22/ min and >50% of radiological involvement of lung with typical lesions.
* FiO2 remain static or improving, along with > 30% deranged ≥ 2 biochemical markers CRP > 20 mg/l, LDH > 600 U/L, D.Dimer > 0.5mg/l or 500 ng/ml, Serum Ferritin < 500 ng/ml or mcg/l will be included in clinical trial.

Exclusion Criteria:

* Heart failure,
* Cardiac arrest
* Decompensated liver cirrhosis,
* Decompensated psychiatric disorder
* Contraindication for corticosteroids
* Leukopenia <1000/mm or neutropenia <500/mm
* Recent or history of bone marrow or solid organ transplantation

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2020-05-01 (Actual); Primary Completion 2020-12-30 (Estimated); Study Completion 2020-12-30 (Estimated)

PRIMARY OUTCOMES:
Clinical response after administration | 10 days
  Clinical improvement of COVID-19 patients by methylprednisolone.

SECONDARY OUTCOMES:
Clinical response to treatment | 28 days
  Overall survival of COVID-19 patients after drug administration.
Duration of hospitalization | 28 days
  Number of days of hospital admission either in ICU or HDUs till date of discharge

CONTACTS AND LOCATIONS:
Overall Officials: Sardar Al-Fareed Zafar, FCPS, Study Director — Post-Graduate Medical Institute, Lahore General Hospital, Lahore Pakistan
Locations (1):
- Muhammad Irfan Malik, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wang Y, Jiang W, He Q, Wang C, Wang B, Zhou P, Dong N, Tong Q. A retrospective cohort study of methylprednisolone therapy in severe patients with COVID-19 pneumonia. Signal Transduct Target Ther. 2020 Apr 28;5(1):57. doi: 10.1038/s41392-020-0158-2. No abstract available. PMID 32341331
- [Background] Xu Z, Shi L, Wang Y, Zhang J, Huang L, Zhang C, Liu S, Zhao P, Liu H, Zhu L, Tai Y, Bai C, Gao T, Song J, Xia P, Dong J, Zhao J, Wang FS. Pathological findings of COVID-19 associated with acute respiratory distress syndrome. Lancet Respir Med. 2020 Apr;8(4):420-422. doi: 10.1016/S2213-2600(20)30076-X. Epub 2020 Feb 18. No abstract available. PMID 32085846
- [Background] Huang C, Wang Y, Li X, Ren L, Zhao J, Hu Y, Zhang L, Fan G, Xu J, Gu X, Cheng Z, Yu T, Xia J, Wei Y, Wu W, Xie X, Yin W, Li H, Liu M, Xiao Y, Gao H, Guo L, Xie J, Wang G, Jiang R, Gao Z, Jin Q, Wang J, Cao B. Clinical features of patients infected with 2019 novel coronavirus in Wuhan, China. Lancet. 2020 Feb 15;395(10223):497-506. doi: 10.1016/S0140-6736(20)30183-5. Epub 2020 Jan 24. PMID 31986264